CLINICAL TRIAL: NCT04363177
Title: Mental Health of Urban Mothers (MUM) Study: A Multi-center Randomized Controlled Trial
Brief Title: Global Mental Health of Urban Mothers
Acronym: MUM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Principal Investigator, Simone Eliane, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P2SKP3_187728
Record Dates: First submitted 2020-04-21; First posted 2020-04-27 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Perinatal Depression; COVID19; Anxiety; PTSD; Pregnancy Related
MeSH Terms: conditions — COVID-19; Anxiety Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-based psychosocial peer-to-peer support (Experimental): Web-based psychosocial peer-to-peer support, using "Thinking Healthy" two times during pregnancy
  Interventions: Behavioral: Web-based psychosocial peer-to-peer support
- Standard perinatal care (Active Comparator): Perinatal standard care in Hong Kong, Shanghai
  Interventions: Behavioral: Web-based psychosocial peer-to-peer support

INTERVENTIONS:
Behavioral: Web-based psychosocial peer-to-peer support — The evidence-based eHealth peer-to-peer psychosocial intervention "Thinking Healthy", will be tested in this RCT. In line with the World Health Organization's mhGAP Intervention Guide (mhGAP-IG), "Thinking Healthy" is used to identify and manage perinatal mental health conditions (distress, symptoms of depression, and anxiety) in non-specialized psychosocial support setting.

SUMMARY:
Mental health disorders are common during pregnancy and the postnatal period, and can have serious adverse effects on the well-being of woman and child. Every tenth woman has depressive symptoms and 5% suffer major depression during pregnancy. The consequences for global mental health due to the novel coronavirus disease, COVID-19, are likely to be significant and may have long-term impact on the global burden of disease. Pregnant women may be particularly vulnerable due to partial immune suppression. Besides physical vulnerability, the women could be at increased risk of mental health problems, such as anxiety, depression, and post-traumatic stress disorder (PTSD), due to social distancing leading to less support from the family and friends, and in some cases, partners not being allowed to be present during prenatal visits, labor and delivery. Furthermore, many pregnant women may feel insecure and worried about the effect of COVID-19 on their unborn child, if the women get infected during pregnancy. Today, young urban women are used to utilizing internet services frequently and efficiently. Therefore, providing mental health support to pregnant women via web-based support may be effective in ameliorating their anxiety/depression and reduce the risk of serious mental health disorders leading to improved maternal and perinatal outcomes.

DETAILED DESCRIPTION:
Pregnancy is a period of transition and great change, which may make some women more vulnerable to mental health problems. It is known that depressive symptoms during pregnancy may influence birth outcomes. Perinatal mental health disorders may become more prevalent during a time of acute crisis, and the prevalence of maternal anxiety, distress, and perinatal depression can be expected to increase globally, as a result of the COVID-19 pandemic. However, there might be cross-national differences in the risk factors and impact of pandemic on the prevalence of perinatal mental health disorders.

Some pregnant women might be predisposed to posttraumatic stress disorder (PTSD) during a crisis situation, such as the COVID-19 pandemic. Mothers who developed PTSD in response to the 9/11 terrorist attacks had lower morning and evening salivary cortisol levels, compared to mothers who did not develop PTSD. Beyond effects on the mother alone, perinatal mental health issues can have long-term effects on child´s mental and physical health, as well as the participants behavior and cognition. Distress in pregnant women may affect the fetus and is known to induce epigenetic changes in the placental genes. Increased risk of psychopathology is observed in children exposed to maternal prenatal distress. Elevated maternal cortisol and epigenetic regulation of placental glucocorticoid-pathway genes are potential mechanisms for these observations. Women often express feelings of inadequacy in the new mothering role, which can furthermore negatively impact the participants mental health and the relationship to the infant.

Effective treatments are needed to address high global rates of postpartum depression (PPD) with onset typically within 4 weeks after delivery and maternal depression up to two years after delivery. Programs aimed at reducing PPD could achieve the most cost-efficient results by focusing efforts in the critical time periods around childbirth. Web-based psychosocial support provided by trained public health nurses is an effective treatment method for PPD. Limited public health resources are challenges to the accessibility of mental health services, which is why the use of web-based psychosocial support could be a good alternative. Women perceive the risk for themselves or their infants to be above average during global crises, which increases the levels of uncertainty. However, face-to-face consultations during a pandemic are likely to increase the risk of disease transmission. Therefore, easily accessible eHealth support could provide fast and resource-effective care during the COVID-19 pandemic.

The study will generate evidence on whether web-based early intervention programs could be efficient in ameliorating the risk and severity of perinatal mental health disorders, and inform best clinical practice for women affected by the consequences of the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 12 and 18 weeks of gestation
* Viable intrauterine pregnancy.

Exclusion Criteria:

* History of severe psychiatric
* Substance abuse disorder
* Requiring medical treatment
* Presence of fetal chromosomal/structural abnormality

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale (EPDS) | 4-6 weeks postpartum
  To investigate the impact of a web-based psychosocial intervention on Edinburgh Postnatal Depression Scale (EPDS) in urban women living in Hong Kong and Shanghainese women.
  Scores of EPDS range from min = 0 to max=30. The higher the score, the more depressed a woman is.

SECONDARY OUTCOMES:
Mental health status and COVID-19 | 4-6 weeks postpartum
  Correlation between mental health status (EPDS, GAD7, IES-R) and COVID-19 pandemic among pregnant women.
  GAD 7 Generalized anxiety questionnaire IES-R Impact Event Scale to assess Post traumatic stress Disorder (PTSD) COVID-19 questionnaire
Socio-economic status (education level, income, marital status, profession, nationality) | 4-6 weeks postpartum
  Impact of web-based psychosocial intervention on mental health and pregnancy outcomes among women from different socio-economic and cultural environments.
  Socio-economic information gained by sociodemographic questions.
Elective CS | 4-6 weeks postpartum
  Relationship between mental health status of pregnant women and rates of elective cesarean section (CS) on maternal request.

CONTACTS AND LOCATIONS:
Overall Officials: Simone E Schwank, PhD, Principal Investigator — Karolinska Institute CLINTEC; Ganesh Acharya, MD PhD, Study Director — Karolinska Institute CLINTEC
Locations (2):
- Shanghai Women's and Children's Health Center, Shanghai, Shanghai Municipality, China
- Chinese University Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brand SR, Engel SM, Canfield RL, Yehuda R. The effect of maternal PTSD following in utero trauma exposure on behavior and temperament in the 9-month-old infant. Ann N Y Acad Sci. 2006 Jul;1071:454-8. doi: 10.1196/annals.1364.041. PMID 16891597
- [Background] Buss C, Davis EP, Hobel CJ, Sandman CA. Maternal pregnancy-specific anxiety is associated with child executive function at 6-9 years age. Stress. 2011 Nov;14(6):665-76. doi: 10.3109/10253890.2011.623250. PMID 21995526
- [Background] Doyle C, Werner E, Feng T, Lee S, Altemus M, Isler JR, Monk C. Pregnancy distress gets under fetal skin: Maternal ambulatory assessment & sex differences in prenatal development. Dev Psychobiol. 2015 Jul;57(5):607-25. doi: 10.1002/dev.21317. Epub 2015 May 6. PMID 25945698
- [Background] Liang H, Acharya G. Novel corona virus disease (COVID-19) in pregnancy: What clinical recommendations to follow? Acta Obstet Gynecol Scand. 2020 Apr;99(4):439-442. doi: 10.1111/aogs.13836. Epub 2020 Mar 5. No abstract available. PMID 32141062
- [Background] Thapa SB, Mainali A, Schwank SE, Acharya G. Maternal mental health in the time of the COVID-19 pandemic. Acta Obstet Gynecol Scand. 2020 Jul;99(7):817-818. doi: 10.1111/aogs.13894. No abstract available. PMID 32374420
- [Background] Monk C, Feng T, Lee S, Krupska I, Champagne FA, Tycko B. Distress During Pregnancy: Epigenetic Regulation of Placenta Glucocorticoid-Related Genes and Fetal Neurobehavior. Am J Psychiatry. 2016 Jul 1;173(7):705-13. doi: 10.1176/appi.ajp.2015.15091171. Epub 2016 Mar 25. PMID 27013342
- [Background] Brummelte S, Galea LA. Postpartum depression: Etiology, treatment and consequences for maternal care. Horm Behav. 2016 Jan;77:153-66. doi: 10.1016/j.yhbeh.2015.08.008. Epub 2015 Aug 28. PMID 26319224
- [Derived] Schwank SE, Chung HF, Hsu M, Fu SC, Du L, Zhu L, Huang HY, Andersson E, Acharya G. Mental health of Urban Mothers (MUM) study: a multicentre randomised controlled trial, study protocol. BMJ Open. 2020 Nov 27;10(11):e041133. doi: 10.1136/bmjopen-2020-041133. PMID 33247023